CLINICAL TRIAL: NCT02422082
Title: The Effect of Lactobacillus Reuteri ATCC PTA 6475 on Volumetric Bone Mineral Density in Patients With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Mattias Lorentzon, Professor, Specialist physician, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRvBMD
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Osteopenia
Keywords: Osteopenia; Lactobacillus reuteri; Volumetric bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri (Active Comparator): Lactobacillus reuteri (L. reuteri) ATCC PTA 6475 at a dose of 5 000 000 000 CFU as a powder in a stick-pack, orally twice daily (morning and evening) yielding a total daily dose of 10 000 000 000 CFU per day, for 12 months.
  Interventions: Dietary Supplement: L. reuteri
- Placebo (Placebo Comparator): Placebo product identical to the active product (L. reuteri) in taste and appearance but without the active component, orally twice daily, for 12 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri — Dietary supplementation with L. reuteri twice daily for 12 months
  Other Names: Lactobacillus reuteri ATCC PTA 6475
  Arms: L. reuteri
Dietary Supplement: Placebo — Dietary supplementation with placebo twice daily for 12 months
  Arms: Placebo

SUMMARY:
Lactobacillus reuteri (L. reuteri) has been widely studied in clinical trials and has probiotic, health-promoting effects in both adults and children, and is safe for human consumption. Animal models indicate that treatment with L. reuteri has positive effects on bone metabolism and bone density. In other animal models of diabetes and the metabolic syndrome, positive effects on blood glucose and weight have been reported. The present double-blind, placebo-controlled, randomized study is designed to investigate if dietary supplementation with L. reuteri twice daily for 12 months has any effect on bone density, body composition, inflammation, or metabolic and endocrine markers in elderly women with osteopenia.

DETAILED DESCRIPTION:
The role of the gut microbes for human health has gained considerable interest in recent years. Lactobacillus reuteri (L.reuteri) is a naturally occurring bacterial species in the human gut. L. reuteri has been widely studied in clinical trials of adults and children and treatment with L. reuteri is safe and is associated with health-promoting effects in humans. In animal models, L. reuteri has anti-inflammatory effects and in ovariectomized mice supplementation with L. reuteri partly prevented the bone loss induced by estrogen deficiency. Furthermore, both bone density and bone formation increased in male mice in another mice model. In mice with medically induced diabetes mellitus, L. reuteri reduced blood glucose and in a mouse model mimicking the metabolic syndrome, L. reuteri prevented diet-induced obesity. The present study is a double-blind, placebo-controlled, randomized, study in 90 elderly women with osteopenia recruited from the population. These women will be treated with L. reuteri or placebo orally twice daily for 12 months. The effects on bone will be investigated with dual energy x-ray absorptiometry, high-resolution peripheral quantitative computed tomography, and bone turnover markers. Hormones and markers of inflammation and metabolism will be followed as well as changes in the gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* bone mineral density T-score less than -1 but more than -2.5 in the total hip or femoral neck or lumbar spine (L1-L4) by dual energy x-ray absorptiometry
* signed informed consent
* stated availability throughout the entire study period
* mental ability to understand and willingness to fulfill all the details of the protocol

Exclusion Criteria:

* untreated hyperthyroidism
* rheumatoid arthritis
* diagnosed with disease causing secondary osteoporosis within the last year, including primary hyperparathyroidism, chronic obstructive pulmonary disease, inflammatory bowel disease, celiac disease, or diabetes
* recently diagnosed malignancy (within the last 5 years)
* per oral corticosteroid use
* use of antiresorptive therapy, including systemic hormone replacement therapy, bisphosphonates, strontium ran elate
* use of teriparatide (current or during the last 3 years)
* participation in other clinical interventional trials
* use of antibiotics within 2 months preceding the inclusion

Ages: 75 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Total tibia volumetric bone mineral density | 12 months
  Change in percent in total tibia volumetric bone mineral density compared to placebo group after 1 year of dietary supplementation with L. reuteri

SECONDARY OUTCOMES:
Trabecular volumetric bone mineral density | 12 months
  Change in percent in trabecular volumetric bone mineral density compared to placebo group after 1 year of dietary supplementation with L. reuteri
Cortical volumetric bone mineral density | 12 months
  Change in percent in cortical volumetric bone mineral density compared to placebo group after 1 year of dietary supplementation with L. reuteri
Cortical thickness | 12 months
  Change in percent in cortical thickness compared to placebo group after 1 year of dietary supplementation with L. reuteri
Cortical porosity | 12 months
  Change in percent in cortical porosity compared to placebo group after 1 year of dietary supplementation with L. reuteri
Areal bone mineral density | 12 months
  Change in percent in areal bone mineral density compared to placebo group after 1 year of dietary supplementation with L. reuteri
Bone material strength index | 12 months
  Change in percent in bone material strength index compared to placebo group after 1 year of dietary supplementation with L. reuteri
Blood pressure | 12 months
  Change in percent in blood pressure compared to placebo group after 1 year of dietary supplementation with L. reuteri
Change in gut microbiota composition | 3-12 months
  Change in percent in gut microbiota composition compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Ultrasensitive C-reactive protein | 3-12 months
  Change in percent in ultrasensitive C-reactive protein in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Interleukin-10 | 3-12 months
  Change in percent in interleukin-10 in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Interleukin-17 | 3-12 months
  Change in percent in interleukin-17 in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Tumor-necrosis factor-alpha | 3-12 months
  Change in percent in tumor-necrosis factor-alpha in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Tartrate-resistent alkaline phosphatase 5b | 3-12 months
  Change in percent in tartrate-resistent alkaline phosphatase 5b in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Cross-linked N-terminal telopeptide | 3-12 months
  Change in percent in cross-linked N-terminal telopeptide in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Bone-specific alkaline phosphatase | 3-12 months
  Change in percent in bone-specific alkaline phosphatase in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Receptor activator of nuclear factor kappa B (RANK) | 3-12 months
  Change in percent in RANK in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Receptor activator of nuclear factor kappa B ligand (RANK-ligand) | 3-12 months
  Change in percent in RANK-ligand in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Osteocalcin | 3-12 months
  Change in percent in osteocalcin in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Blood glucose | 3-12 months
  Change in percent in blood glucose compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Haemoglobin A1C | 3-12 months
  Change in percent in haemoglobin A1C compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Apolipoprotein A1 (ApoA1) | 3-12 months
  Change in percent in ApoA1 compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Apolipoprotein B (ApoB) | 3-12 months
  Change in percent in ApoB compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Cholesterol | 3-12 months
  Change in percent in cholesterol compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
High density lipoprotein (HDL) | 3-12 months
  Change in percent in HDL compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Low density lipoprotein (LDL) | 3-12 months
  Change in percent in LDL compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Triglycerides | 3-12 months
  Change in percent in triglycerides compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Oxytocin | 3-12 months
  Change in percent in oxytocin in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Estradiol | 3-12 months
  Change in percent in estradiol in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Leptin | 3-12 months
  Change in percent in leptin in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Adiponectin | 3-12 months
  Change in percent in adiponectin in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Testosterone | 3-12 months
  Change in percent in testosterone in serum compared to placebo after 3, 6, 9, and 12 months of dietary supplementation with L. reuteri
Lean mass | 12 months
  Change in percent in lean mass compared to placebo after 12 months of dietary supplementation with L. reuteri
Fat mass | 12 months
  Change in percent in fat mass compared to placebo after 12 months of dietary supplementation with L. reuteri

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Lorentzon, MD, PhD, Principal Investigator — Dept Geriatrics, Sahlgrenska University Hospital
Locations (1):
- Geriatric Medicine, Mölndal Hospital, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams MR, Marteau P. On the safety of lactic acid bacteria from food. Int J Food Microbiol. 1995 Oct;27(2-3):263-4. doi: 10.1016/0168-1605(95)00067-t. No abstract available. PMID 8579995
- [Background] Reid G, Kim SO, Kohler GA. Selecting, testing and understanding probiotic microorganisms. FEMS Immunol Med Microbiol. 2006 Mar;46(2):149-57. doi: 10.1111/j.1574-695X.2005.00026.x. PMID 16487295
- [Background] Britton RA, Irwin R, Quach D, Schaefer L, Zhang J, Lee T, Parameswaran N, McCabe LR. Probiotic L. reuteri treatment prevents bone loss in a menopausal ovariectomized mouse model. J Cell Physiol. 2014 Nov;229(11):1822-30. doi: 10.1002/jcp.24636. PMID 24677054
- [Background] McCabe LR, Irwin R, Schaefer L, Britton RA. Probiotic use decreases intestinal inflammation and increases bone density in healthy male but not female mice. J Cell Physiol. 2013 Aug;228(8):1793-8. doi: 10.1002/jcp.24340. PMID 23389860
- [Background] Fak F, Backhed F. Lactobacillus reuteri prevents diet-induced obesity, but not atherosclerosis, in a strain dependent fashion in Apoe-/- mice. PLoS One. 2012;7(10):e46837. doi: 10.1371/journal.pone.0046837. Epub 2012 Oct 9. PMID 23056479